CLINICAL TRIAL: NCT02703987
Title: A Randomized, Controlled, Double-blind, Cross-over, Single-centre Study to Investigate the Effect of a Fermented Infant Formula on Lactose Digestion in Lactose Intolerant Adults
Brief Title: HYBRID: Hydrogen Breath Test in Lactose Digestion
Acronym: HYBRID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Dig.1.C.I/0
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): Fermented infant milk formula
  Interventions: Other: Fermented infant milk formula
- Group II (Active Comparator): Non-fermented infant milk formula
  Interventions: Other: Non-fermented infant milk formula

INTERVENTIONS:
Other: Fermented infant milk formula
  Arms: Group I
Other: Non-fermented infant milk formula
  Arms: Group II

SUMMARY:
The purpose of this study is to investigate the effect of a fermented infant formula on lactose digestion in lactose intolerant adults.

ELIGIBILITY:
Inclusion Criteria:

BMI between 18.5 and 24.9 kg/m2 inclusive Lactose intolerant

The following criteria need to be checked at visit 2:

* Lactose intolerance confirmed by positive Hydrogen Breath Test (HBT) (i.e. if there are two or more samples with hydrogen level > 20 ppm increase compared to baseline sample between 90 mins and 240 min sampling time point).
* At least one sample with hydrogen level > 20 ppm increase compared to baseline between 90 mins and 180 mins sampling time point.

Exclusion Criteria:

History of gastrointestinal disorders Current illness which could interfere with the study (e.g. diarrhea, regurgitation) Any history of cow's milk protein allergy or known allergy to galacto-oligosaccharides Any current participation or within 8 weeks of study start, in any other study involving investigational or marketed products, any medical procedures, or any surgical methods.

Any antibiotic, laxative or colonic cleansing treatments within 4 weeks of study start Any administration of probiotic in the 1 week prior to study start Investigator's uncertainty about willingness or ability of subject to comply with protocol requirements

The following criteria need to be checked at visit 2:

* Level of hydrogen > 20 ppm in the baseline breath sample.
* An early peak of hydrogen (i.e. hydrogen level > 20 ppm increase compared to baseline value) in the first 60 minutes after ingestion of the study products.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ngai Moh Law, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were terminated before randomisation (1 due to sponsor decision to withdraw, and 1 due to consent withdrawal).
Groups:
- Sequence 1 (Test at Visit 3 Followed by Control at Visit 4): Test product: 35g of Gallia Lactofidus 1 + 11.2g lactose to match an oral load of 20g lactose, 250mL (reconstituted), once as breakfast, had to be consumed within 10 mins
  Control product: 35g of Nursie 1 + 10g maltodextrin to match an oral load of 20g lactose and the carbohydrate load as test product, 250mL (reconstituted), once as breakfast, had to be consumed within 10 mins.
- Sequence 2 (Control at Visit 3 Followed by Test at Visit 4): Control product: 35g of Nursie 1 + 10g maltodextrin to match an oral load of 20g lactose and the carbohydrate load as test product, 250mL (reconstituted), once as breakfast, had to be consumed within 10
  Test product: 35g of Gallia Lactofidus 1 + 11.2g lactose to match an oral load of 20g lactose, 250mL (reconstituted), once as breakfast, had to be consumed within 10 mins
Period: Visit 3 Intervention (1 Day)
Arm/Group | Sequence 1 (Test at Visit 3 Followed by Control at Visit 4) | Sequence 2 (Control at Visit 3 Followed by Test at Visit 4)
Started | 14 | 14
Completed | 13 | 11
Not Completed | 1 | 3
Period: Washout (Minimum 5 Days)
Arm/Group | Sequence 1 (Test at Visit 3 Followed by Control at Visit 4) | Sequence 2 (Control at Visit 3 Followed by Test at Visit 4)
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0
Period: Visit 4 Intervention (1 Day)
Arm/Group | Sequence 1 (Test at Visit 3 Followed by Control at Visit 4) | Sequence 2 (Control at Visit 3 Followed by Test at Visit 4)
Started | 13 | 11
Completed | 12 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Test at visit 3, Control at visit 4
- Sequence 2: Control at visit 3, Test at visit 4
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (6.5) | 30.6 (4.6) | 30.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 13 | 12 | 25
  Indian | 0 | 1 | 1
  Malay | 0 | 1 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Log of First Postprandial Peak Change of Hydrogen Concentration
Description: This is measured as the log of the first change >20ppm peak value compared to baseline between 90 minutes and 240 minutes. If there was no change >20ppm at all between 90 minutes and 240 minutes, it is the maximum change compared to baseline in that interval
Time Frame: Postprandial peak hydrogen in breath within 4 hours after ingestion of study product; samples taken at 30 minute intervals for 4 hours, i.e. at 90, 120, 150, 180, 210 and 240 minutes at Visits 3 and 4
Population: At Visit 3, 14 subjects took the control product and at Visit 4, 13 subjects took the control product. Therefore, 27 subjects took the control product in total.
  At Visit 3, 14 subjects took the test product and at Visit 4, 11 subjects took the test product. Therefore, 25 subjects took the test product in total.
Measure: Least Squares Mean (Standard Error); unit: log(ppm)
Groups:
- Control: Non-fermented infant milk formula
- Test: Fermented infant milk formula
Arm/Group | Control | Test
Number analyzed (Participants) | 27 | 25
log(ppm)
  Baseline | 1.21 (0.10) | 1.10 (0.10)
  Post-baseline | 3.38 (0.08) | 3.59 (0.09)
Statistical Analysis 1: Comparison: Control vs Test; Test type: Superiority; p = 0.0801, Mixed Models Analysis; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.04 to 0.67], Standard Error of Mean 0.17

2. Primary Outcome: Log of Maximum Postprandial Change in Hydrogen Concentration
Description: This is measured as the maximum change in postprandial hydrogen concentration (ppm) compared to baseline between 90 minutes and 240 minutes
Time Frame: Maximum postprandial hydrogen in breath within 4 hours after ingestion of study product; samples taken at 30 minute intervals for 4 hours, i.e. at 90, 120, 150, 180, 210 and 240 minutes at Visits 3 and 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: log(ppm)
Arm/Group | Control | Test
Number analyzed (Participants) | 27 | 25
log(ppm)
  Baseline | 1.21 (0.10) | 1.09 (0.11)
  Post-baseline | 3.70 (0.10) | 3.93 (0.11)
Statistical Analysis 1: Comparison: Control vs Test; Test type: Superiority; p = 0.0714, Mixed Models Analysis; Mean Difference (Net) = 0.34, 95% CI 2-sided [-0.03 to 0.71], Standard Error of Mean 0.18

3. Secondary Outcome: Square Root of Postprandial Incremental Area Under Curve (iAUC) of Hydrogen Concentration From 30 Minutes to 240 Minutes
Description: The iAUC of hydrogen concentration from 30 to 240 minute sampling time points is calculated with the triangular rule (reference: Wolever TM. Effect of blood sampling schedule and method of calculating the area under the curve on validity and precision of glycaemic index values. Br J Nutr. 2004 Feb;91(2):295-301). The square root of the iAUC is then taken for the outcome measure
Time Frame: Hydrogen in breath within 4 hours after ingestion of study product; samples taken at 30 minute intervals for 4 hours, i.e. at 30, 60, 90, 120, 150, 180, 210 and 240 minutes at Visits 3 and 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: sqrt(ppm*min)
Arm/Group | Control | Test
Number analyzed (Participants) | 27 | 25
sqrt(ppm*min) | 66.22 (4.42) | 75.78 (4.59)
Statistical Analysis 1: Comparison: Control vs Test; Test type: Superiority; p = 0.0609, Mixed Models Analysis; Mean Difference (Net) = 9.56, 95% CI 2-sided [-0.48 to 19.6], Standard Error of Mean 4.85

ADVERSE EVENTS:
Time Frame: From visit 1 (day -14 to 0) to visit 4 (day 11 to 15)
Description: Adverse events were collected throughout the study period and were documented by Investigator at Visit 2 (Day 1), Visit 3 (Day 6-8), and Visit 4 (Day 11-15).
Arm/Group | Control | Test
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 26/27 | 25/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=27) | Test (N=25)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 4 (4) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Defecation Urgency (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 14 (14)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 15 (16) | 16 (16)
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 9 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results communication be submitted to Nutricia Research for review and comment prior to publication at least sixty (60) days prior to submission for publication, public dissemination, or review by a publication committee.

All reasonable comments made by Nutricia Research in relation to a proposed publication by Contractor will be incorporated into the publication.